CLINICAL TRIAL: NCT00579098
Title: Atorvastatin for Prevention of Atrial Fibrillation Recurrence Following Pulmonary Veins Isolation: A Double-Blind, Placebo-Controlled, Randomized Pilot Trial
Brief Title: The Use of Statins Following a Left Atrial Catheter Ablation Procedure to Prevent Atrial Fibrillation
Acronym: ATTAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Paul A. Friedman, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-005460
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation; Arrhythmia; Inflammation; Endothelial Dysfunction
Keywords: Atrial Fibrillation; Arrhythmia; Pulmonary Vein Isolation; Left atrial catheter ablation; Inflammation; Endothelial dysfunction
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): Lipitor (atorvastatin) 80 mg tablet taken once daily by mouth for 90 days
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo (dummy) tablet taken once daily by mouth for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg tablet taken by mouth daily for 90 days
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — Placebo tablet taken by mouth once daily for 90 days
  Other Names: Placebo (dummy) tablet to match appearance of atorvastatin
  Arms: Placebo

SUMMARY:
To investigate whether statin therapy utilizing the drug Lipitor (atorvastatin) might be effective in preventing short-and long-term atrial fibrillation (AF) following a left atrial ablation procedure. We further hypothesize this reduction will result from diminished peri-procedural inflammation, which will be reflected in lower C-Reactive Protein (CRP) values in the blood.

DETAILED DESCRIPTION:
Although pharmacologic therapy is the traditional mainstay of therapy for AF, curative therapy has recently become possible.

There is growing evidence that inflammation may be involved in the pathogenesis of AF. CRP, a sensitive marker of systemic inflammation, is increased in patients with AF compared with patients in sinus rhythm. Elevated CRP levels are associated with increased likelihood of new onset AF and with recurrence of AF after successful cardioversion. Clinical and basic laboratory evidence suggests that, in addition to being potent lipid-lowering agents, statins may also have anti-inflammatory properties and protective effect against AF.

125 eligible patients with AF, undergoing left atrial ablation, will be randomly assigned in a 1:1 ratio to receive daily 80 mg of atorvastatin or placebo in a double-blind fashion for 3 months after their ablation procedure.

Patients will have baseline lipids, CRP, endothelial function tests and Quality of Life (QoL) surveys compared with testing at 3 months post ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = to 18 years of age
* Clinically indicated left atrial ablation procedure for atrial fibrillation

Exclusion Criteria:

* Known malignancy
* Known inflammatory disease
* Surgery or trauma or myocardial infarction in the previous month
* Known contraindication to statin therapy
* Elevated liver enzymes above two times the upper limit of normal
* Patients already receiving therapy with any statin, niacin or fibrates at the time of their randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Friedman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Aviles RJ, Martin DO, Apperson-Hansen C, Houghtaling PL, Rautaharju P, Kronmal RA, Tracy RP, Van Wagoner DR, Psaty BM, Lauer MS, Chung MK. Inflammation as a risk factor for atrial fibrillation. Circulation. 2003 Dec 16;108(24):3006-10. doi: 10.1161/01.CIR.0000103131.70301.4F. Epub 2003 Nov 17. PMID 14623805
- [Background] Malouf JF, Kanagala R, Al Atawi FO, Rosales AG, Davison DE, Murali NS, Tsang TS, Chandrasekaran K, Ammash NM, Friedman PA, Somers VK. High sensitivity C-reactive protein: a novel predictor for recurrence of atrial fibrillation after successful cardioversion. J Am Coll Cardiol. 2005 Oct 4;46(7):1284-7. doi: 10.1016/j.jacc.2005.06.053. PMID 16198844
- [Background] Patti G, Chello M, Candura D, Pasceri V, D'Ambrosio A, Covino E, Di Sciascio G. Randomized trial of atorvastatin for reduction of postoperative atrial fibrillation in patients undergoing cardiac surgery: results of the ARMYDA-3 (Atorvastatin for Reduction of MYocardial Dysrhythmia After cardiac surgery) study. Circulation. 2006 Oct 3;114(14):1455-61. doi: 10.1161/CIRCULATIONAHA.106.621763. Epub 2006 Sep 25. PMID 17000910
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Result] Suleiman M, Koestler C, Lerman A, Lopez-Jimenez F, Herges R, Hodge D, Bradley D, Cha YM, Brady PA, Munger TM, Asirvatham SJ, Packer DL, Friedman PA. Atorvastatin for prevention of atrial fibrillation recurrence following pulmonary vein isolation: a double-blind, placebo-controlled, randomized trial. Heart Rhythm. 2012 Feb;9(2):172-8. doi: 10.1016/j.hrthm.2011.09.016. Epub 2011 Sep 13. PMID 21920481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in this trial between January 2008 and December 2009 at Mayo Clinic in Rochester, Minnesota (USA).
Pre-assignment Details: 847 patients were screened and of those, 567 were excluded, primarily because they were already receiving statin therapy (68%) and/or had known inflammatory disease (16%). 280 met entry criteria but 155 were not willing to participate. 125 were enrolled in the study.
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 62 | 63
Completed | 53 | 55
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — AF returned after ablation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10) | 57 (10) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  United States | 62 | 63 | 125
Paroxysmal Atrial Fibrillation [Number; unit: Participants] — Paroxysmal atrial fibrillation is atrial fibrillation that comes and goes, starting and stopping suddenly. Not all patients experience this type of atrial fibrillation, therefore, the number reported for each group will differ from the number of overall participants per group.
  Participants | 44 | 46 | 90
Duration of Atrial Fibrillation [Median (Full Range); unit: Months] | 4 [1 to 24] | 4 [1 to 18] | 4 [1 to 24]
Years of Atrial Fibrillation [Mean (Standard Deviation); unit: Years] | 5.7 (4.90) | 4.9 (3.96) | 5.3 (4.45)
Concomitant Conditions [Number; unit: Participants] — Not all subjects had all concomitant medical conditions, therefore the number reported for each condition will not match the overall/total number of subjects per treatment group.
  Participants
    Hypertension | 20 | 16 | 36
    Diabetes Mellitus | 1 | 0 | 1
    Coronary Artery Disease | 0 | 0 | 0
    Congestive Heart Failure | 0 | 3 | 3
    Dilated cardiomyopathy | 1 | 0 | 1
    Hypertrophic cardiomyopathy | 0 | 0 | 0
    Valvular heart disease | 6 | 5 | 11
    Old Cardiovascular Accident/Transient Ischemic Att | 0 | 0 | 0
    Chronic kidney disease | 1 | 2 | 3
    Chronic lung disease | 1 | 2 | 3
    Sleep apnea | 14 | 12 | 26
Medication on admission [Number; unit: Participants] — Not all subjects were taking all medications upon admission, therefore the number reported for each medication class will not match the overall/total number of subjects per treatment group.
  Participants
    Aspirin | 28 | 30 | 58
    Oral anticoagulation | 46 | 41 | 87
    Beta blocker | 35 | 30 | 65
    ACE inhibitors/Angiotensin Receptor Blockers | 12 | 7 | 19
Antiarrhythmic drugs [Number; unit: Participants] — Not all subjects were taking antiarrhythmic drugs upon admission, therefore the numbers reported will differ from the number of overall subjects in each treatment group.
  Participants
    Total on any antiarrhythmic drug | 28 | 33 | 61
    Sotalol/dofetilide | 14 | 9 | 23
    Amiodarone | 1 | 4 | 5
    Sodium Channel Blocker Class IC | 13 | 20 | 33
Echocardiographic parameter-LA diameter, long axis [Mean (Standard Deviation); unit: millimeters] — LA = left atrium (chamber of heart)
  millimeters | 58.4 (6.7) | 57.5 (7.7) | 57.9 (7.2)
Echocardiographic parameter-LA volume index [Mean (Standard Deviation); unit: cc/m^2] | 40.4 (0.7) | 39.4 (13.1) | 39.9 (13.8)
Echocardiographic parameter-LVEF [Mean (Standard Deviation); unit: Percentage] — LVEF= left ventricular ejection fraction, which is the volume of blood pumped out of the heart with each heartbeat. A normal LVEF ranges from 55-70%. A LVEF of 65, for example, means that 65% of the total amount of blood in the left ventricle is pumped out with each heartbeat.
  Percentage | 60 (10) | 60 (9) | 60 (10)
Procedural time [Mean (Standard Deviation); unit: Minutes] | 110 (39) | 113 (47) | 111 (42)
Anatomical area of ablation [Number; unit: Participants] — The catheter ablation procedure involves intentional destruction of left atrial (LA) tissue via radiofrequency energy and is used to treat atrial fibrillation (AF). Lesions often extend to the pericardium and pericardiac tissues, therefore the total number of various anatomical ablation locations reported will not total the overall number of subjects in a treatment group.
  Participants
    Wide-area circumferential ablation | 44 | 46 | 90
    LA isthmus | 12 | 7 | 19
    Roof line | 12 | 8 | 20
    Cavotricuspid isthmus line | 49 | 51 | 100
    Nonpulmonary vein foci | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Without Symptoms of Atrial Fibrillation at 3 Months
Description: Asymptomatic recurrence was defined as any atrial arrhythmia lasting more than 30 seconds. This was assessed by an electrocardiogram (ECG) and 72-hour Holter monitor recordings. At the end of the study, 336 ECG and Holter recordings were available for analysis (172 in the atorvastatin group and 164 in the placebo group).
Time Frame: Baseline through 3 months
Population: Intent-to-treat analysis population.
Measure: Number; unit: Percentage of subjects
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 62 | 63
Percentage of subjects | 95 | 93.5
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = 0.75, Log Rank — A p-value of < 0.05 was considered statistically significant

2. Secondary Outcome: Percentage of Subjects Without Atrial Arrhythmia at 3 Months
Description: Percentage of subjects without atrial arrhythmia (as opposed to atrial fibrillation) recurrence, irrespective of symptoms. Atrial arrhythmias included AF, atrial tachycardia and atrial flutter.
Time Frame: Baseline through 3 months
Population: Intent-to-treat analysis population.
Measure: Number; unit: Percentage of subjects
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 62 | 63
Percentage of subjects | 85 | 88
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = 0.37, Log Rank — A p-value of < 0.05 was considered statistically significant

3. Secondary Outcome: Change in Mean C-Reactive Protein Level
Time Frame: Baseline and 3 months
Population: Intent-to-treat analysis population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 62 | 63
mg/dL | -0.75 (3) | 2.1 (19.9)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = 0.11, t-test, 2 sided — A p-value of < 0.05 was considered statistically significant

4. Secondary Outcome: Change in Mean Quality of Life Score
Description: A visual analogue scale (VAS) was used to collect the subject's perception of their current state of health/quality of life. The VAS consists of a vertical 20 centimeter scored line (like a thermometer) with the ends labelled best imaginable health state at the top (100) and worst imaginable health state at the bottom (0). The subject marked a single line to grade his/her own current level of function at the baseline visit and again at the 3 month visit. The average change in VAS score from baseline to 3 months later is reported for each treatment group.
Time Frame: Baseline and 3 months
Population: Intent-to-treat analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 62 | 63
units on a scale | 13 (18) | 11 (18)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = 0.53, t-test, 2 sided — Comparison between treatment groups. A p-value of < 0.05 was considered statistically significant

5. Secondary Outcome: Change in Lipid Levels
Description: The change from baseline to 3 months in blood cholesterol levels (total cholesterol, LDL or low-density lipoprotein and HDL or high-density lipoprotein) was calculated.
Time Frame: Baseline and 3 months
Population: Intent-to-treat analysis population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 62 | 63
mg/dL
  Change in total cholesterol | -50 (42) | 15 (29)
  Change in LDL (low-density lipoprotein) cholestero | -47 (35) | 9 (23)
  Change in HDL (high-density lipoprotein) cholest. | 3 (7) | 3 (9)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; The change in total cholesterol was compared between treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — A p-value of < 0.05 was considered statistically significant
Statistical Analysis 2: Comparison: Atorvastatin vs Placebo; The change in LDL cholesterol was compared between treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — A p-value of < 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Atorvastatin vs Placebo; The change in HDL cholesterol was compared between treatment groups; Test type: Superiority or Other; p = 0.92, t-test, 2 sided — A p-value of < 0.05 was considered statistically significant

ADVERSE EVENTS:
Time Frame: Baseline to 3 months post ablation procedure.
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 1/62 | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=62) | Placebo (N=63)
Clot formation in left atrium during ablation procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Puncture of the subclavian artery during ablation procedure (Surgical and medical procedures) | 1 (1) | 0 (0) — The puncture was repaired surgically.
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Pain resolved two days after stopping Lipitor.
Elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0) — Headache resolved within 24 hours of stopping atorvastatin.
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The population was restricted to patients who did not have an indication for statin treatment. The lack of transtelephonic or prolonged Holter monitoring likely resulted in underestimation of the rate of asymptomatic episodes of AF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No